CLINICAL TRIAL: NCT01043380
Title: Plaque REgression With Cholesterol Absorption Inhibitor or Synthesis Inhibitor Evaluated by IntraVascular UltraSound
Acronym: PRECISE-IVUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kumamoto University (Other)
Responsible Party: Principal Investigator, Hisao Ogawa, Professor, Kumamoto University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMIN000002959
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Hypercholesterolemia; Coronary Artery Disease
Keywords: Heart Diseases; Hyperlipidemia; Atorvastatin; Ezetimibe; Cardiovascular Diseases; Hypercholesterolemia; Coronary Artery Disease; Dyslipidemias; Intravascular Ultrasound
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease; Heart Diseases; Hyperlipidemias; Cardiovascular Diseases; Dyslipidemias | interventions — Combined Modality Therapy; Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LZ group (Experimental)
  Interventions: Drug: Combination therapy with Lipitor [Atorvastatin] and Zetia [Ezetimibe]
- L group (Active Comparator)
  Interventions: Drug: Lipitor (Atorvastatin) monotherapy

INTERVENTIONS:
Drug: Combination therapy with Lipitor [Atorvastatin] and Zetia [Ezetimibe] — Zetia 10 mg/dl + Lipitor. The dosage of Lipitor will be titrated up to a maximum of 20 mg/day with a treatment goal of lowering LDL-C below 70 mg/dl.
  Arms: LZ group
Drug: Lipitor (Atorvastatin) monotherapy — The dosage will be titrated up to a maximum of 20 mg/day, which is the highest approved regimen by the Ministry of Health, Labor and Welfare of Japan, with a treatment goal of lowering LDL-C below 70 mg/dl.
  Arms: L group

SUMMARY:
The purpose of this study was to evaluate the difference in the effect of coronary plaque regression (as measured by intravascular ultrasound [IVUS] imaging) between cholesterol absorption inhibitor and cholesterol synthesis inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent,
* 30 to 85 years old,
* Plan to undergo PCI and LDL-C >= 100 mg/dL

Exclusion Criteria:

* Familial hypercholesterolemia
* Being treated with Zetia (Ezetimibe)
* Being treated with Fibrates
* Renal insufficiency (serum creatinine >= 2.0 mg/dl)
* Altered hepatic function (serum aspartate aminotransferase or alanine aminotransferase >= 3-folds of standard value in each institute)
* Undergoing hemodialysis or peritoneal dialysis
* Allergic to Lipitor and/or Zetia
* Severe underlying disease
* Lack of decision-making capacity
* Recognized as inadequate by attending doctor

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2010-01; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to follow-up in percent atheroma volume (PAV) in the target lesion | before randomization & 9-12 months after randomization

SECONDARY OUTCOMES:
Percentage change from baseline (before randomization) to follow-up (9-12 months after randomization) in the atheroma volume | before randomization & 9-12 months after randomization
Change and percentage change from baseline to follow-up in the minimum lumen diameter (MLD) and percent diameter stenosis (%DS) | before randomization & 9-12 months after randomization
Percentage changes from baseline to follow-up in serum lipids | before randomization & 9-12 months after randomization
Correlation between regression of coronary plaque and serum lipids profiles | before randomization & 9-12 months after randomization
Changes in hs-CRP from baseline to follow-up | before randomization & 9-12 months after randomization
Correlation between regression of coronary plaque and inflammatory markers (white blood cell count and hs-CRP) | before randomization & 9-12 months after randomization
Change and percentage change from baseline to follow-up in the PV of the PCI target lesion | before randomization & 9-12 months after randomization
Change and percentage change from baseline to follow-up in the MLD and %DS of the PCI target lesion | before randomization & 9-12 months after randomization
MACE (cardiac death, non-fatal Q wave and/or non-Q wave myocardial infarction, target vessel revascularization [percutaneous coronary intervention or coronary artery bypass grafting]) | before randomization & 9-12 months after randomization
All-cause death | before randomization & 9-12 months after randomization
Safety (Adverse events, subjective symptoms/objective findings, physical tests), blood tests [hematology, clinical chemistry, glucose metabolism test], urinalysis) | before randomization & 9-12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, MD, PhD, Study Chair — Kumamoto University, Graduate School of Medical Sciences
Locations (1):
- Kumamoto University, Kumamoto, Japan

REFERENCES:
- [Derived] Fujisue K, Nagamatsu S, Shimomura H, Yamashita T, Nakao K, Nakamura S, Ishihara M, Matsui K, Yamamoto N, Koide S, Matsumura T, Fujimoto K, Tsunoda R, Morikami Y, Matsuyama K, Oshima S, Sakamoto K, Izumiya Y, Kaikita K, Hokimoto S, Ogawa H, Tsujita K. Impact of statin-ezetimibe combination on coronary atheroma plaque in patients with and without chronic kidney disease - Sub-analysis of PRECISE-IVUS trial. Int J Cardiol. 2018 Oct 1;268:23-26. doi: 10.1016/j.ijcard.2018.04.051. Epub 2018 Jun 18. PMID 29925472
- [Derived] Tsujita K, Yamanaga K, Komura N, Sakamoto K, Sugiyama S, Sumida H, Shimomura H, Yamashita T, Oka H, Nakao K, Nakamura S, Ishihara M, Matsui K, Sakaino N, Nakamura N, Yamamoto N, Koide S, Matsumura T, Fujimoto K, Tsunoda R, Morikami Y, Matsuyama K, Oshima S, Kaikita K, Hokimoto S, Ogawa H; PRECISE-IVUS Investigators. Lipid profile associated with coronary plaque regression in patients with acute coronary syndrome: Subanalysis of PRECISE-IVUS trial. Atherosclerosis. 2016 Aug;251:367-372. doi: 10.1016/j.atherosclerosis.2016.05.025. Epub 2016 May 20. PMID 27318866
- [Derived] Tsujita K, Sugiyama S, Sumida H, Shimomura H, Yamashita T, Yamanaga K, Komura N, Sakamoto K, Oka H, Nakao K, Nakamura S, Ishihara M, Matsui K, Sakaino N, Nakamura N, Yamamoto N, Koide S, Matsumura T, Fujimoto K, Tsunoda R, Morikami Y, Matsuyama K, Oshima S, Kaikita K, Hokimoto S, Ogawa H; PRECISE-IVUS Investigators. Impact of Dual Lipid-Lowering Strategy With Ezetimibe and Atorvastatin on Coronary Plaque Regression in Patients With Percutaneous Coronary Intervention: The Multicenter Randomized Controlled PRECISE-IVUS Trial. J Am Coll Cardiol. 2015 Aug 4;66(5):495-507. doi: 10.1016/j.jacc.2015.05.065. PMID 26227186